CLINICAL TRIAL: NCT03665311
Title: Saline Versus Albumin Fluid for Extracorporeal Removal With Slow Low Efficiency Dialysis (SAFER-SLED): A Feasibility Study
Brief Title: Saline Versus Albumin Fluid for Extracorporeal Removal With Slow Low Efficiency Dialysis Feasibility Study
Acronym: SAFER-SLED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRRF 316
Record Dates: First submitted 2018-07-19; First posted 2018-09-11 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Renal Replacement Therapy; Acute Kidney Injury; Hypotension
Keywords: Albumin; Normal Saline; Dialysis; Intensive Care Unit
MeSH Terms: conditions — Acute Kidney Injury; Hypotension | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two parallel arms 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The packaging for normal saline and 25% albumin will be identical (glass bottles) and be covered. The intravenous tubing will have an opaque sleeve to mask any colour discrepancy in the 2 products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Placebo Comparator): 100 mL 0.9% Normal Saline at the initiation of SLED and another 100 mL 0.9% Normal Saline after 4 hours of treatment
  Interventions: Other: Normal Saline
- 25% Albumin fluid (Active Comparator): 100 mL 25% Albumin fluid at the initiation of SLED and another 100 mL 25% Albumin fluid after 4 hours of treatment
  Interventions: Biological: 25% Albumin fluid

INTERVENTIONS:
Biological: 25% Albumin fluid — 25% Albumin fluid (100 mL)
  Arms: 25% Albumin fluid
Other: Normal Saline — 0.9% Normal Saline (100 mL)
  Arms: Normal Saline

SUMMARY:
Objective: The primary aim of this 60 patient feasibility trial is to determine if, for critically ill patients treated with SLED for AKI, randomization to receive albumin (25%) boluses versus normal saline placebo boluses is feasible, with respect to the recruitment rate, blinding and adherence to the protocol.

DETAILED DESCRIPTION:
Background: Intravenous albumin (25%) boluses are frequently given to critically ill patients during slow low-efficiency dialysis (SLED) treatments for acute kidney injury (AKI). The intention of giving albumin during SLED is to stabilize the blood pressure to permit more aggressive overall fluid removal with ultrafiltration; however, there is little evidence to support this expensive practice.

Objective: The primary aim of this feasibility trial is to determine if, for critically ill patients treated with SLED for AKI, randomization to receive albumin (25%) boluses versus normal saline placebo boluses is feasible, with respect to the recruitment rate, blinding and adherence to the protocol.

The results of this feasibility trial will help us to plan and carry out a multicentre pilot trial comparing the efficacy of the interventions in achieving fluid removal in critically ill patients with AKI on SLED.

Design: A randomized controlled trial with two parallel arms. Setting: The mixed medical-surgical intensive care units of a Canadian tertiary care hospital.

Study Population: 60 patients with AKI requiring treatment with SLED (by definition, Kidney Disease Improving Global Outcomes (KDIGO) stage 3 AKI). Intervention: Participants will be randomized to receive either albumin (25%) boluses or normal saline placebo boluses during their SLED treatments.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 yrs;
2. AKI treated with SLED (stage 3 AKI per Kidney Disease Improving Global Outcomes (KDIGO) AKI guidelines48).

Exclusion Criteria:

1. SLED initiated for non AKI-related indication (i.e. concurrent intoxication; treatment of hypothermia);
2. receiving chronic dialysis treatments;
3. history of allergic reaction to albumin;
4. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 24 months
  Percentage of eligible patients that are successfully recruited into the study

SECONDARY OUTCOMES:
Adherence to intervention | Through study completion, on average 1 year.
  Percentage of SLED sessions in which patients received their allocated intervention (or placebo).
Completeness of follow-up | 24 months
  Percentage of patients who have complete data available with respect to the primary and other secondary outcomes at the end of the study.
Volume removal achieved during SLED sessions | Through study completion, on average 1 year.
  Overall fluid removal (i.e. percentage of target ultrafiltration achieved)calculated as the actual ultrafiltration volume divided by the target (ordered) ultrafiltration volume).
New or increased vasopressor use during SLED sessions | Through study completion, on average 1 year.
  Initiation or any increase in vasopressor dose(s) before the completion of a SLED session relative to the start.
Change in mean arterial blood pressure (MAP) < 55 mmHg during SLED sessions | Through study completion, on average 1 year.
  Percentage of SLED sessions during which patients' MAP (defined as [(2X diastolic blood pressure) + systolic blood pressure]/3) falls to <55 mmHg at any time during the SLED session.
Change in MAP of >=20 mmHg during the SLED sessions. | Through study completion, on average 1 year.
  Percentage of SLED sessions during which patients' MAP falls by >=20 mmHg relative to their MAP at the start of the SLED session.

CONTACTS AND LOCATIONS:
Overall Officials: Edward G Clark, MD, MSc, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Clark EG, McIntyre L, Watpool I, Kong JWY, Ramsay T, Sabri E, Canney M, Hundemer GL, Brown PA, Sood MM, Hiremath S. Intravenous albumin for the prevention of hemodynamic instability during sustained low-efficiency dialysis: a randomized controlled feasibility trial (The SAFER-SLED Study). Ann Intensive Care. 2021 Dec 13;11(1):174. doi: 10.1186/s13613-021-00962-x. PMID 34902089
- [Derived] Clark EG, McIntyre L, Ramsay T, Tinmouth A, Knoll G, Brown PA, Watpool I, Porteous R, Montroy K, Harris S, Kong J, Hiremath S. Saline versus albumin fluid for extracorporeal removal with slow low-efficiency dialysis (SAFER-SLED): study protocol for a pilot trial. Pilot Feasibility Stud. 2019 May 30;5:72. doi: 10.1186/s40814-019-0460-3. eCollection 2019. PMID 31161046